CLINICAL TRIAL: NCT01246960
Title: Randomized, Placebo-Controlled, Double-Blind Phase 2 Study of mFOLFOX6 Chemotherapy Plus Ramucirumab Drug Product(IMC-1121B) Versus mFOLFOX6 Plus Placebo for Advanced Adenocarcinoma of the Esophagus, Gastroesophageal Junction or Stomach
Brief Title: A Study of Ramucirumab in Participants With Gastric, Esophageal, and Gastroesophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14057; I4T-MC-JVBT (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-08; First posted 2010-11-24 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Stomach Cancer; Esophageal Cancer
Keywords: cancer; stomach; esophagus; gastroesophageal
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasms | interventions — Ramucirumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramucirumab (Experimental): * Oxaliplatin 85 milligrams per square meter (mg/m^2) given on Day 1 of a 2-week cycle
  * Leucovorin 400 mg/m^2 given on Day 1 of a 2-week cycle
  * 5-Fluorouracil (5-FU) 400 mg/m^2 bolus given on Day 1 of a 2-week cycle
  * 5-FU 2400 mg/m^2 continuously given over 46-48 hours on Day 1 of a 2-week cycle
  * Ramucirumab 8 milligrams per kilogram (mg/kg) given on Day 1 of a 2-week cycle
  Participants will receive study treatment every 2 weeks until disease progression, unacceptable toxicity, or another withdrawal criterion is met
  Interventions: Biological: Ramucirumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil
- Placebo (Placebo Comparator): * Oxaliplatin 85 mg/m^2 given on Day 1 of a 2-week cycle
  * Leucovorin 400 mg/m^2 given on Day 1 of a 2-week cycle
  * 5-FU 400 mg/m^2 bolus given on Day 1 of a 2-week cycle
  * 5-FU 2400 mg/m^2 continuously given over 46-48 hours on Day 1 of a 2-week cycle
  * Placebo given on Day 1 of a 2-week cycle
  Participants will receive study treatment every 2 weeks until disease progression, unacceptable toxicity, or another withdrawal criterion is met
  Interventions: Drug: Placebo; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil

INTERVENTIONS:
Biological: Ramucirumab — Administered intravenously
  Other Names: LY3009806; IMC-1121B
  Arms: Ramucirumab
Drug: Placebo — Administered intravenously
  Arms: Placebo
Drug: Oxaliplatin — Administered intravenously
Drug: Leucovorin — Administered intravenously
Drug: 5-Fluorouracil — Administered intravenously
  Other Names: 5-FU

SUMMARY:
The purpose of this study is to determine whether ramucirumab when used in conjunction with chemotherapy treatment can help participants with stomach, esophagus, and gastroesophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of adenocarcinoma of the esophagus, gastroesophageal junction (GEJ), or stomach
* Metastatic or locally advanced, unresectable disease at time of study entry
* Provided signed informed consent and is amenable to compliance with protocol schedules and testing
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1 at study entry
* Adequate renal, hematological, and hepatic function
* Measurable or non-measurable disease at the time of study entry
* Resolution to Grade less than or equal to 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0, of all clinically significant toxic effects of prior locoregional therapy, surgery, or other anticancer therapy, except where otherwise mentioned in the eligibility criteria
* Eligible participants of reproductive potential (both sexes) must agree to use adequate contraceptive methods (hormonal or barrier methods) during the study period and at least 12 weeks after the last dose of study therapy
* Life expectancy of greater than or equal to 3 months
* Willingness to provide blood and tissue samples for research purposes. Submission of tumor specimen is mandatory for participation in this study, if a histologic, paraffin-embedded specimen exists (either from a surgical resection or biopsy); submission of paraffin block or a minimum of 8 unstained slides is required if sufficient sample. NOTE: If insufficient additional tissue exists (that is, all tissue has been utilized for prior diagnostic purposes), participation in the study is allowable without the requirement for an additional biopsy; this situation must be discussed with the study principal investigator and/or the ImClone medical monitor or designee.

Exclusion Criteria:

* The participant has received prior first-line systemic therapy for advanced/unresectable and/or metastatic disease (prior adjuvant or neo-adjuvant therapy is permitted)
* Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to study entry
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the participant ineligible for entry into this study
* The participant is receiving chronic therapy with nonsteroidal anti-inflammatory agents (NSAIDs; for example, indomethacin, ibuprofen, naproxen, or similar agents) or other antiplatelet agents (for example, clopidogrel, ticlopidine, dipyridamole, anagrelide). Aspirin use at doses up to 325 milligrams per day (mg/day) is permitted.
* The participant has significant third-space fluid retention (for example, ascites or pleural effusion), and is not amenable for required repeated drainage
* The participant is pregnant or breastfeeding
* Uncontrolled intercurrent illness including, but not limited to, active or uncontrolled clinically serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled thromboembolic, or hemorrhagic disorder, psychiatric illness/social situations, or other co-morbid systemic illnesses, or other severe concurrent disease
* Immunocompromised participants including participants known to be human immunodeficiency virus (HIV) positive.
* Progressive disease less than or equal to 12 months of completing platinum or 5-FU treatment, including capecitabine, if given previously in the perioperative (adjuvant or neoadjuvant) setting
* Current or recent (within 28 days prior to randomization) treatment with an investigational drug that has not received regulatory approval for any indication at the time of study entry, or participation in another interventional clinical trial. Participants participating in surveys or observational studies are eligible to participate in this study.
* Are currently enrolled in, or discontinued within the last 28 days from, a clinical trial involving ramucirumab drug product (DP), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Received prior therapy with an antiangiogenic agent (including but not limited to bevacizumab, sunitinib, or sorafenib)
* Major surgical procedure or significant traumatic injury less than 28 days prior to randomization, or anticipation of need for elective or planned major surgical procedure during the course of the study. Subcutaneous venous access device placement within 7 days prior to randomization
* Clinically significant peripheral neuropathy at the time of registration
* Known central nervous system metastases that are symptomatic or untreated
* New York Heart Association (NYHA) classification III-IV congestive heart failure
* Greater than normal risk of bleeding or coagulopathy in the absence of therapeutic anticoagulation; Grade 3/4 gastrointestinal bleeding within 3 months prior to registration; active bleeding (that is, within 14 days prior to first dose of study therapy); or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices)
* Participant has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, stroke, transient ischemic attack (TIA), cerebrovascular accident, or unstable angina, less than or equal to 6 months prior to registration
* Clinically significant vascular disease (for example, aortic aneurysm, aortic dissection) for which more than minimal intervention is being administered or planned
* History of hypertensive crisis or hypertensive encephalopathy or current poorly-controlled hypertension despite standard medical management
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess less than 6 months prior to registration
* Known hypersensitivity to any of the treatment components of modified FOLFOX6 (mFOLFOX6) (oxaliplatin, 5-FU, and leucovorin) or ramucirumab DP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (58):
- United States (58):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anchorage, Alaska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alhambra, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redondo Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Junction, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Englewood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewiston, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Louis Park, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bozeman, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hackensack, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunmore, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spartanburg, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kirkland, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Vernon, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Wisconsin

REFERENCES:
- [Derived] Yoon HH, Bendell JC, Braiteh FS, Firdaus I, Philip PA, Cohn AL, Lewis N, Anderson DM, Arrowsmith E, Schwartz JD, Gao L, Hsu Y, Xu Y, Ferry D, Alberts SR, Wainberg ZA. Ramucirumab combined with FOLFOX as front-line therapy for advanced esophageal, gastroesophageal junction, or gastric adenocarcinoma: a randomized, double-blind, multicenter Phase II trial. Ann Oncol. 2016 Dec;27(12):2196-2203. doi: 10.1093/annonc/mdw423. Epub 2016 Oct 20. PMID 27765757

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramucirumab and mFOLFOX6: Ramucirumab: 8 milligrams per kilogram (mg/kg) intravenous infusion administered on Day 1 of each cycle (14 days/cycle). In Cycles 1 and 2, there was a 1-hour observation prior to administering modified FOLFOX6 (mFOLFOX6).
  mFOLFOX6: Administered intravenously per manufacturer's instructions for each drug substance on Day 1 of each cycle (14 days/cycle).
  * Oxaliplatin 85 milligrams per square meter (mg/m^2)
  * Leucovorin 400 mg/m^2
  * 5-Fluorouracil (5-FU) 400 mg/m^2 bolus
  * 5-FU 2400 mg/m^2 continuous given over 46-48 hours
  Participants received study treatment every 2 weeks until disease progression, unacceptable toxicity, or another withdrawal criterion was met.
- Placebo and mFOLFOX6: Placebo: intravenous infusion administered on Day 1 of each cycle (14 days/cycle). In Cycles 1 and 2, there was a 1-hour observation prior to administering mFOLFOX6.
  mFOLFOX6: Administered intravenously per manufacturer's instructions for each drug substance on Day 1 of each cycle (14 days/cycle).
  * Oxaliplatin 85 mg/m^2
  * Leucovorin 400 mg/m^2
  * 5-FU 400 mg/m^2 bolus
  * 5-FU 2400 mg/m^2 continuous given over 46-48 hours
  Participants received study treatment every 2 weeks until disease progression, unacceptable toxicity, or another withdrawal criterion was met.
Period: Overall Study
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Started | 84 | 84
Received Any Quantity of Study Drug | 82 | 80
Completed | 78 | 80
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal (by participant or physician) | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all randomized participants.
Groups:
- Ramucirumab and mFOLFOX6: Ramucirumab: 8 mg/kg intravenous infusion administered on Day 1 of each cycle (14 days/cycle). In Cycles 1 and 2, there was a 1-hour observation prior to administering mFOLFOX6.
  mFOLFOX6: Administered intravenously per manufacturer's instructions for each drug substance on Day 1 of each cycle (14 days/cycle).
  * Oxaliplatin: 85 mg/m^2
  * Leucovorin: 400 mg/m^2
  * 5-FU: 400 mg/m^2 bolus
  * 5-FU: 2400 mg/m^2 continuous given over 46-48 hours
  Participants received study treatment every 2 weeks until disease progression, unacceptable toxicity, or another withdrawal criterion was met.
- Placebo and mFOLFOX6: Placebo: intravenous infusion administered on Day 1 of each cycle (14 days/cycle). In Cycles 1 and 2, there was a 1-hour observation prior to administering mFOLFOX6.
  mFOLFOX6: Administered intravenously per manufacturer's instructions for each drug substance on Day 1 of each cycle (14 days/cycle).
  * Oxaliplatin: 85 mg/m^2
  * Leucovorin: 400 mg/m^2
  * 5-FU: 400 mg/m^2 bolus
  * 5-FU: 2400 mg/m^2 continuous given over 46-48 hours
  Participants received study treatment every 2 weeks until disease progression, unacceptable toxicity, or another withdrawal criterion was met.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6 | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 56 | 98
  >=65 years | 42 | 28 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 63 | 61 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 80 | 75 | 155
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 3 | 3 | 6
  White | 77 | 76 | 153
Region of Enrollment [Number; unit: participants]
  United States | 84 | 84 | 168

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined using Response Evaluation Criteria in Solid Tumors [RECIST version (v.) 1.1] as the time from randomization to the first observation of progressive disease (PD) or death due to any cause, whichever came first. PD was a ≥20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of ≥5 millimeters (mm); the appearance of ≥1 new lesions or unequivocal progression of non-target lesions. If a participant did not have a baseline disease assessment, PFS time was censored at the randomization date, regardless of whether or not PD or death was observed. Participants not known to have died or have objective PD were censored at the last post-baseline radiological assessment date.
Time Frame: Randomization to measured PD or date of death from any cause (up to Month 25.0)
Population: ITT population: all randomized participants. Fourteen participants in the Ramucirumab and mFOLFOX6 treatment arm and 15 participants in the Placebo and mFOLFOX6 treatment arm were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 84 | 84
months | 6.4 [5.8 to 9.3] | 6.7 [5.6 to 7.8]
Statistical Analysis 1: Comparison: Ramucirumab and mFOLFOX6 vs Placebo and mFOLFOX6; Test type: Superiority or Other; p = 0.886, Stratified Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.69 to 1.37]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS was censored at the date of the last follow-up visit for participants who were alive or lost to follow-up.
Time Frame: Randomization to date of death from any cause (up to Month 28.3)
Population: ITT population: all randomized participants. Twenty-seven participants in the Ramucirumab and mFOLFOX6 treatment arm and 32 participants in the Placebo and mFOLFOX6 treatment arm were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 84 | 84
months | 11.7 [10.2 to 14.6] | 11.5 [9.0 to 15.3]
Statistical Analysis 1: Comparison: Ramucirumab and mFOLFOX6 vs Placebo and mFOLFOX6; Test type: Superiority or Other; p = 0.712, Stratified Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.73 to 1.58]

3. Secondary Outcome: Percentage of Participants Achieving an Objective Response (Objective Response Rate)
Description: The percentage of participants who achieved a best overall response of partial response (PR) or complete response (CR) is reported. Response was defined using RECIST, v. 1.1 criteria. CR was the disappearance of all lesions and pathological lymph node reduction in the short axis to <10 mm. PR was a ≥30% decrease in the sum of the diameters of target lesions. The percentage of participants with objective response=(number of participants whose best overall response achieved was CR or PR/number of participants treated)*100.
Time Frame: Randomization to measured PD (up to Month 23.0)
Population: ITT population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 84 | 84
percentage of participants | 45.2 [34.3 to 56.5] | 46.4 [35.5 to 57.6]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined using RECIST v. 1.1 criteria as the time from the date criteria were met for the first objectively recorded CR or PR until the first date criteria for PD were met or death from any cause. CR was the disappearance of all lesions and pathological lymph node reduction in the short axis to <10 mm. PR was a ≥30% decrease in the sum of the diameters of target lesions. PD was a ≥20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of ≥5 mm; the appearance of ≥1 new lesions or unequivocal progression of non-target lesions. Participants who were not known to have died and who did not have PD were censored at the date of the last tumor assessment prior to the date of any subsequent systemic anticancer therapy.
Time Frame: Time of first response to measured PD (up to Month 23.0)
Population: Randomized participants who achieved an objective response of CR or PR. Eight participants in the Ramucirumab and mFOLFOX6 treatment arm and 8 participants in the Placebo and mFOLFOX6 treatment arm were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 38 | 39
months | 7.4 [4.2 to 8.4] | 5.8 [4.4 to 8.0]

5. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP was defined using RECIST v. 1.1 as the time from study randomization to the first date of PD. PD was a ≥20% increase in the sum of the diameters of target lesions with the sum demonstrating an absolute increase of ≥5 mm; the appearance of ≥1 new lesions or unequivocal progression of non-target lesions. TTP was censored at the date of last adequate tumor assessment if death was due to causes other than PD.
Time Frame: Randomization to measured PD (up to Month 25.0)
Population: ITT population: all randomized participants. Thirty-five participants in the Ramucirumab and mFOLFOX6 treatment arm and 31 participants in the Placebo and mFOLFOX6 treatment arm were censored.
Measure: Median (Full Range); unit: months
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 84 | 84
months | 8.7 [6.0 to 9.8] | 7.1 [5.8 to 9.2]
Statistical Analysis 1: Comparison: Ramucirumab and mFOLFOX6 vs Placebo and mFOLFOX6; Test type: Superiority or Other; p = 0.516, Stratified Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.59 to 1.30]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Ramucirumab Antibodies
Description: Participants with treatment-emergent anti-ramucirumab antibodies were participants with a 4-fold increase (2 dilution increase) in immunogenicity titer over baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20).
Time Frame: Months 1, 2, 4, 6, and 8
Population: Randomized participants who received any quantity of ramucirumab or placebo, and were evaluated for the presence of anti-ramucirumab antibodies.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 81 | 77
participants | 0 | 1

7. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: Reported are the number of participants who had ramucirumab/placebo-related: AEs, serious AEs (SAEs), AEs based on common terminology criteria for adverse events (CTCAE) ≥Grade 3, AEs = CTCAE Grade 5, as well as, AEs leading to treatment discontinuation and AEs resulting in death. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion (up to Month 28.3)
Population: Safety population: randomized participants who received any quantity of study drug (Ramucirumab, mFOLFOX6, or placebo).
Measure: Number; unit: participants
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Number analyzed (Participants) | 82 | 80
participants
  Any Ramucirumab/Placebo-Related AE | 64 | 64
  Any Ramucirumab/Placebo-Related SAE | 10 | 12
  Any Ramucirumab/Placebo-Related ≥Grade 3 AE | 36 | 33
  Any Ramucirumab/Placebo-Related Grade 5 AE | 0 | 3
  Any AE Leading to Treatment Discontinuation | 18 | 5
  Any AE with Outcome of Death | 5 | 2

ADVERSE EVENTS:
Arm/Group | Ramucirumab and mFOLFOX6 | Placebo and mFOLFOX6
Serious Adverse Events (participants affected / at risk) | 48/82 | 32/80
Other Adverse Events (participants affected / at risk) | 82/82 | 79/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and mFOLFOX6 (N=82) | Placebo and mFOLFOX6 (N=80)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Device dislocation (General disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 1 (1) | 3 (3)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and mFOLFOX6 (N=82) | Placebo and mFOLFOX6 (N=80)
Anaemia (Blood and lymphatic system disorders) | 29 (41) | 38 (58)
Leukopenia (Blood and lymphatic system disorders) | 7 (18) | 9 (14)
Neutropenia (Blood and lymphatic system disorders) | 29 (76) | 33 (108)
Thrombocytopenia (Blood and lymphatic system disorders) | 30 (62) | 20 (45)
Vision blurred (Eye disorders) | 3 (3) | 6 (7)
Abdominal distension (Gastrointestinal disorders) | 8 (9) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 17 (20) | 14 (20)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10) | 8 (11)
Ascites (Gastrointestinal disorders) | 5 (8) | 2 (2)
Constipation (Gastrointestinal disorders) | 36 (41) | 32 (41)
Diarrhoea (Gastrointestinal disorders) | 36 (67) | 33 (56)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 7 (9) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 10 (15) | 13 (18)
Flatulence (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (9) | 5 (11)
Nausea (Gastrointestinal disorders) | 52 (72) | 56 (82)
Oral pain (Gastrointestinal disorders) | 5 (6) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 10 (16) | 16 (21)
Vomiting (Gastrointestinal disorders) | 32 (49) | 28 (42)
Asthenia (General disorders) | 12 (13) | 8 (13)
Chest pain (General disorders) | 2 (2) | 7 (11)
Chills (General disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 57 (91) | 56 (81)
Mucosal inflammation (General disorders) | 17 (23) | 9 (13)
Oedema peripheral (General disorders) | 20 (30) | 14 (19)
Pyrexia (General disorders) | 9 (12) | 11 (11)
Temperature intolerance (General disorders) | 8 (8) | 14 (17)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 5 (6)
Urinary tract infection (Infections and infestations) | 11 (11) | 9 (12)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (14) | 5 (7)
Alanine aminotransferase increased (Investigations) | 5 (6) | 7 (9)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 11 (18)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 15 (24)
Blood creatinine increased (Investigations) | 5 (11) | 1 (1)
Neutrophil count decreased (Investigations) | 16 (50) | 9 (16)
Platelet count decreased (Investigations) | 19 (45) | 12 (24)
Weight decreased (Investigations) | 28 (41) | 21 (31)
White blood cell count decreased (Investigations) | 5 (8) | 6 (8)
Decreased appetite (Metabolism and nutrition disorders) | 37 (47) | 22 (36)
Dehydration (Metabolism and nutrition disorders) | 21 (28) | 12 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (15) | 10 (22)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (15) | 4 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (23) | 8 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (7) | 6 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (13) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 11 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 (14) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (9)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Dizziness (Nervous system disorders) | 19 (22) | 12 (15)
Dysgeusia (Nervous system disorders) | 13 (14) | 14 (15)
Headache (Nervous system disorders) | 18 (24) | 12 (16)
Memory impairment (Nervous system disorders) | 5 (5) | 0 (0)
Paraesthesia (Nervous system disorders) | 8 (10) | 20 (33)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 6 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 44 (68) | 43 (73)
Anxiety (Psychiatric disorders) | 4 (4) | 8 (8)
Depression (Psychiatric disorders) | 7 (7) | 4 (5)
Insomnia (Psychiatric disorders) | 15 (15) | 20 (24)
Dysuria (Renal and urinary disorders) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 15 (18)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (23) | 16 (24)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (28) | 9 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10) | 8 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6)
Hypertension (Vascular disorders) | 30 (41) | 10 (10)
Hypotension (Vascular disorders) | 7 (10) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.